CLINICAL TRIAL: NCT01186640
Title: Phase II Trial of Combined Immunochemotherapy With Fludarabine, Mitoxantrone, Cyclophosphamide and Alemtuzumab (FMC-Alemtuzumab) in Patients With Previously Treated or Untreated T-Prolymphocytic Leukemia
Brief Title: Combined Immunochemotherapy in Patients With T-Prolymphocytic Leukemia (T-PLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); University of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-PLL2; 2008-001421-34 (EudraCT Number)
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2018-05

CONDITIONS: T-cell-prolymphocytic Leukemia
Keywords: T-PLL; Polychemotherapy; Alemtuzumab; Efficacy
MeSH Terms: conditions — Leukemia, Prolymphocytic, T-Cell | interventions — fludarabine; Mitoxantrone; Cyclophosphamide; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCM-A followed by A-maintenance (Experimental): First treatment phase: Chemoimmunotherapy A-FMC maximum 4 cycles. Second treatment phase: Maintenance-treatment with 30mg Alemtuzumab s.c.
  Interventions: Drug: Fludarabine, Mitoxantrone, Cyclophosphamide and Alemtuzumab; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Fludarabine, Mitoxantrone, Cyclophosphamide and Alemtuzumab — I. First treatment phase: Chemoimmunotherapy A-FMC
  Alemtuzumab:
  Cycle 1+2:
  10 mg s.c., days 1-3
  Cycle 3+4:
  CR: 10 mg s.c., days 1-3 PR/SD: 30 mg s.c., days 1-3 Fludarabine: 20 mg/m2 i.v., days 1-3 Mitoxantrone: 6 mg/m2 i.v., day 1 Cyclophosphamide: 200 mg/m2 i.v., days 1-3 Repeat day 29, maximum 4 cycles. II. Second treatment phase: Maintenance-treatment with 30mg Alemtuzumab s.c. The maintenance therapy will start one month after the Final Staging and will be administered monthly during the first six months plus once in month 10 and 13.
  Other Names: Mabcampath; Fludarabine; Endoxan; Novantron
Drug: Alemtuzumab — maintenance with Alemtuzumab following a induction with combined immunochemotherapy consisting of Fludarabine, cyclophosphamide, mitoxantrone and alemtuzumab
  Other Names: Mabcampath

SUMMARY:
Study hypothesis: Simultaneous FMC-Alemtuzumab administration followed by Alemtuzumab maintenance therapy in patients with T-PLL is feasible, safe and efficient.

DETAILED DESCRIPTION:
As the median survival time of patients with T-PLL is less than 12 months, the treatment of T-PLL is a special challenge.

The overall response rates with conventional chemotherapy or Deoxycoformycin were low (about 30% and 40%), with the monoclonal antibody Alemtuzumab response rates of 50% to 70% were achieved, but the duration of the response was short.

In the previous trial (T PLL 1), the efficacy of the FMC regimen (FMC = Fludarabine, Mitoxantrone and Cyclophosphamide) was tested, a preliminary analysis of 16 patients revealed a response rate of more than 60% after FMC-polychemotherapy and 83% after the subsequent administration of Alemtuzumab.

The goal of the T-PLL2-protocol is to assess if the simultaneous administration of FMC-polychemotherapy and Alemtuzumab with a subsequent Alemtuzumab maintenance therapy is capable of improving the remission rate and the disease-free survival time in patients with T-PLL.

ELIGIBILITY:
Inclusion Criteria:

* Untreated patients with T-prolymphocytic leukemia (T-PLL) according to WHO criteria or pretreated patients (max. one previous treatment) with T-PLL
* Age ≥ 18 years
* WHO performance status of 0-2
* Life expectancy > 6 months
* CIRS score >= 6
* Left ventricular ejection fraction ≥50% confirmed by echo-cardiogram performed < 6 months before inclusion to the trial and after the end of a possible anthracycline containing pretreatment
* Adequate liver function as indicated by a total bilirubin, AST and ALT >= 2 the institutional ULN value, unless directly attributable to the T-PLL
* Creatinine clearance >= 70 ml/min calculated according to the formula of Cockcroft and Gault
* Seronegativity for HIV, HBV or HCV confirmed by serological testing within 6 weeks prior to registration
* Willingness of fertile male and female patients to use a highly effective contraceptive method with a Pearl-Index < 1 during and at least six months after the end of the study treatment (e.g. implants, injectables, oral contraceptives in combination with another contraceptive method, some IUDs, sexual abstinence or vasectomised partner)
* Negative serum pregnancy test one week prior to treatment (required for female patients before and <2 years after onset of menopause)
* Patient's written informed consent

Exclusion Criteria:

* Clinically significant auto-immune cytopenia or clinically significant hemolytic anaemia with suspicion of immune origin, even if Coombs test is negative
* Active secondary malignancy requiring treatment (except basal cell carcinoma or tumour curatively treated by surgery)
* Medical condition requiring prolonged use of oral corticosteroids (> 1 month)
* Cerebral dysfunction, legal incapacity
* Any circumstance at the time of study entry that would preclude completion of the study and required follow-up
* Active infection or severe infection (WHO 4th degree) within the last three months before inclusion to the study
* Participation in any other clinical trial during this study
* Known hypersensitivity to any of the study medications (Fludarabine, Cyclophosphamide, Mitoxantrone or Alemtuzumab)
* Patients who have already received more than 60% of the recommended maximum cumulative dose of an anthracycline (Epirubicine, Adriamycine or Mitoxantrone).

This maximum cumulative dose is defined for the individual substances as follows:

* Epirubicin 900 mg/m²
* Daunorubicin 550 mg/m², (or 400 mg/m² if the patient received mediastinal irradiation)
* Adriamycine (Doxorubicine) 550 mg/m²
* Mitoxantrone 200 mg/m²

  * Patients who already received Fludarabine in combination with Cyclophosphamide or Mitoxantrone
  * Patients who received prior treatment with Alemtuzumab alone or in combination with a purine analogue and who did not achieve a PR that lasted at least 6 months
  * Patients who are employees of the Sponsor (University of Cologne) or the study sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Remission Rate | 2 years after trial started
  Efficacy of the FMC therapy and Alemtuzumab Percentage and 95%-confidence-interval of response rates (CR, CRi, nPR, PR, SD and PD) will be provided.

SECONDARY OUTCOMES:
Overall Survival Time | 4 years after start of trial
  OS will be calculated from the patient´s time of recruitment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, Prof. MD, Principal Investigator — German CLL Study Group
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pflug N, Cramer P, Robrecht S, Bahlo J, Westermann A, Fink AM, Schrader A, Mayer P, Oberbeck S, Seiler T, Zenz T, Durig J, Kreuzer KA, Stilgenbauer S, Eichhorst B, Hallek M, Herling M, Hopfinger G. New lessons learned in T-PLL: results from a prospective phase-II trial with fludarabine-mitoxantrone-cyclophosphamide-alemtuzumab induction followed by alemtuzumab maintenance. Leuk Lymphoma. 2019 Mar;60(3):649-657. doi: 10.1080/10428194.2018.1488253. Epub 2018 Sep 20. PMID 30234404